CLINICAL TRIAL: NCT01366287
Title: A Randomized, Open-Label, Single Dose, Crossover Study To Estimate The Relative Oral Bioavailability And Food Effect Of PF-03882845 In Healthy Adult Volunteers
Brief Title: A Study Of PF-03882845 Absorption In Healthy Volunteers Given Orally As Tablet Versus Suspension Formulations And Effect Of Food On Its Absorption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B0171006
Record Dates: First submitted 2011-01-04; First posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Relative bioavailability; food effect; tablet; suspension; single dose; crossover; healthy subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (3S,3aR)-2-(3-chloro-4-cyanophenyl)-3-cyclopentyl-3,3a,4,5-tetrahydro-2H-benzo(g)indazole-7-carboxylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Suspension/fasted (Experimental)
  Interventions: Drug: PF-03882845
- Tablet/fasted (Experimental)
  Interventions: Drug: PF-03882845
- Tablet/fed (Experimental)
  Interventions: Drug: PF-03882845

INTERVENTIONS:
Drug: PF-03882845 — 25 mg of PF-03882845 suspension (75% SDD) will be given as a single oral dose under fasted condition
  Arms: Suspension/fasted
Drug: PF-03882845 — 25 mg PF-03882845 Tablet (75% SDD) will be given as a single oral dose under fasted condition
  Arms: Tablet/fasted
Drug: PF-03882845 — 25 mg PF-03882845 Tablet (75% SDD) will be given as a single oral dose under fed condition
  Arms: Tablet/fed

SUMMARY:
The primary purpose of this study is to estimate the relative bioavailability and food effect of a PF-03882845 tablet as compared to a suspension formulation used in previous clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years,Females must be of non-childbearing potential. Body mass index of 17.5 to 30.5 kg/m2.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Serum potassium >5 mEq/L at screening.
* Impaired kidney function (estimated GFR <60 mL/min/1.73 m2). History of sensitivity to eplerenone, spironolactone, or related compounds.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
PF-03882845 PK: Cmax, AUCinf, AUClast, Tmax, t1/2, as data permit. | predose and post each dose (24, 48 and 96 hour timepoints)
  Post dose is measured at 24, 48 and 96 hours after dose.
Safety: Safety labs, vital signs, ECGs, physical examinations and adverse event monitoring. | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0171006&StudyName=A%20Study%20Of%20PF-03882845%20Absorption%20In%20Healthy%20Volunteers%20Given%20Orally%20As%20Tablet%20Versus%20Suspension%20Formulations%20And%20Effect%20Of%20Food%20On%20It